CLINICAL TRIAL: NCT04405011
Title: Role of Nucleoside Analogue in Preventing Clinical Reactivation of HBV in HCV/HBV Co-infected Patients Receiving DAA Therapy for Chronic Hepatitis C
Brief Title: NUC in Preventing HBV Reactivation in HCV/HBV Co-infected Patients Receiving DAA for CHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 201807069MINB
Record Dates: First submitted 2020-04-17; First posted 2020-05-28 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-05

CONDITIONS: HBV/HCV Co-infection
Keywords: HCV,HBV
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Entecavir 0.5mg daily for 24 weeks (Experimental): Entecavir will be delivered for 24-week and will be the experimental arm
  Interventions: Drug: 24-week Entecavir
- Entecavir 0.5mg daily for 12 weeks (Active Comparator): 12-week entecavir will be served as active comparator
  Interventions: Drug: 12-week Entecavir
- Control (No Intervention): Control group does not receive prophylactic ETV

INTERVENTIONS:
Drug: 24-week Entecavir — Entecavir 0.5mg for 24 weeks will be delivered
  Other Names: Prophylaxis arm 1
  Arms: Entecavir 0.5mg daily for 24 weeks
Drug: 12-week Entecavir — Entecavir for 12 weeks will be delivered and serve as the active comparator arm
  Other Names: Prophylaxis arm 2
  Arms: Entecavir 0.5mg daily for 12 weeks

SUMMARY:
HBV reactivation is common in HCV/HBV coinfected patients receiving DAA therapy for chronic hepatitis C. How to prevent HBV reactivation remains unclear. In this trial, we aim to investigate whether prophylactic nucleos(t)ide analogue (NUC) at the start of DAA could prevent HBV reactivation or not. And whether prolonged NUC prophylaxis (24 weeks) would be better than 12-week prophylaxis. This will be a three-arm, open-label, randomized, active controlled, study. Totally, 60 HBV/HCV co-infected treatment-naïve or treatment-experienced patients without decompensated liver cirrhosis will be included in this study. Group 1 patients (n=20) will receive 12-week ETV from the start of DAA therapy. Group 2 patients (n=20) will receive 24-week ETV from the start of DAA till 12 weeks after end of DAA. Group 3 patients (n=20) will not receive ETV during the period of DAA and will serve as controls. The rate of HBV reactivation and clinical reactivation will be compared among 3 groups of patients. Expected outcomes: The rate of HBV reactivation and clinical reactivation will be lower in the ETV prophylaxis group, and will be the lowest in the group receiving 24-week ETV prophylaxis.

DETAILED DESCRIPTION:
We will determine the incidence of virologic and clinical reactivation of HBV during DAA treatment for CHC, in two prophylactic groups versus control group. We will also examine whether extending the duration of prophylactic NUC would be more beneficial than the 3-month prophylaxis regimen.

Patients with the following criteria will be enrolled: age ≥20 years; anti-HCV positive and HCV RNA >1000 IU/ml; any HCV genotype; all received 12 weeks of DAA treatment; treatment naïve or experienced of pegylated interferon/ribavirin; concurrent HBV infection which is defined by positive HBsAg for at least 6 months. Patients with the following criteria will be excluded: history of treatment regimen that included any kind of direct antiviral agents; presence of other etiology of chronic hepatitis including HIV, autoimmune hepatitis, NASH, etc; uncontrolled diabetes mellitus (Hba1c >8.5); current evidence or suspicion of malignancy; severe cardiovascular or other severe comorbid diseases; autoimmune disorders; presence of liver cirrhosis clinically or pathologically; any one of following hematology or biochemical or clinical abnormalities: AST/ALT >10x ULN, Albumin <3.5g/dL, Bilirubin >2.5mg/dL, eGFR <30 ml/min/1.73m2, prothrombin time prolongation >4 sec or INR >1.7, platelet count <100 x 103 uL, and history or presence of ascites or hepatic encephalopathy; child-bearing age women without the willing to contraceptive control; and pregnant women or lactating women.

Briefly, 60 HCV/HBV coinfected patients will be enrolled and randomized to receive 12-week DAA regimen for reimbursed for the the treatment of patients with CHC in Taiwan.

Entecavir (0.5mg; ETV) 1 # daily will be used in the prophylactic group. Group 1 patients (n=20) will receive 12-week ETV from the start of DAA therapy. Group 2 patients (n=20) will receive 24-week ETV from the start of DAA till 12 weeks after end of DAA. Group 3 patients (n=20) will not receive ETV during the period of DAA and serve as controls. The rate of HBV reactivation and clinical reactivation will be compared among 3 groups of patients.

The primary endpoint will be the incidence of virologic and clinical reactivation of HBV during DAA treatment for CHC. Secondary objectives include the rate of HBV virologic and clinical reactivation between 12-week versus 24-week entecavir (ETV) prophylaxis during and after DAA treatment; the profiles of serum HBV DNA/qHBsAg during and after DAA treatment; and sustained virological response at post-DAA treatment 12 weeks (SVR12).

The data will be expressed as percentages for category variables and as mean +- standard deviation for continuous variables. Category variables will be evaluated by Chi-square test or Fisher exact test. Student's t test or Mann-Whitney U test will be applied for comparison of the continuous variables. Multivariate analysis will be used to identify factors that are associated with HBV reactivation. A p value less than 0.05 is considered to be significant.

ELIGIBILITY:
Inclusion criteria

1. Age ≥20 years;
2. Anti-HCV positive and HCV RNA >1000 IU/ml;
3. Any HCV genotype; all received 12 weeks of DAA treatment.
4. Treatment naïve or experienced of pegylated interferon/ribavirin;
5. Concurrent HBV infection which is defined by positive HBsAg for at least 6 months.

Exclusion criteria

1. History of treatment regimen that included any kind of direct antiviral agents;
2. Presence of other etiology of chronic hepatitis including HIV, autoimmune hepatitis, NASH, etc;
3. Uncontrolled diabetes mellitus (Hba1c >8.5);
4. Current evidence or suspicion of malignancy;
5. Severe cardiovascular or other severe comorbid diseases;
6. Autoimmune disorders;
7. Presence of liver cirrhosis clinically or pathologically;
8. Any one of following hematology or biochemical or clinical abnormalities:

   AST/ALT >10x ULN, Albumin <3.5g/dL, Bilirubin >2.5mg/dL, eGFR <30 ml/min/1.73m2, prothrombin time prolongation >4 sec or INR >1.7, platelet count <100 x 103 uL, and history or presence of ascites or hepatic encephalopathy.
9. Child-bearing age women without the willing to contraceptive control; pregnant women or lactating women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-28 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
HBV virologic and clinical reactivation rates | 72 weeks
  The primary endpoint will be the incidence of virologic and clinical reactivation of HBV during DAA treatment for CHC.

SECONDARY OUTCOMES:
HBV reactivation rate: 12-week prophylaxis versus 24-week prophylaxis | 72 weeks
  12 weeks or 24 weeks of ETV prophylaxis in the control of HBV activity during and after DAA treatment
Profiles of serum HBV DNA/qHBsAg during and after DAA treatment. | 72 weeks
  The profiles of HBV DNA and qHBsAg will be compared among 3 study groups
Sustained virological response at post-DAA treatment 12 weeks (SVR12) | 72 weeks
  The SVR12 will be compared among 3 study groups

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Jen Liu, MDPHD, Principal Investigator — Department of Internal Medicine, NTUH
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - TC Chen, Taipei

REFERENCES:
- [Derived] Cheng PN, Liu CJ, Chen CY, Tseng KC, Lo CC, Peng CY, Lin CL, Chiu HC, Chiu YC, Chen PJ. Entecavir Prevents HBV Reactivation During Direct Acting Antivirals for HCV/HBV Dual Infection: A Randomized Trial. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2800-2808. doi: 10.1016/j.cgh.2021.11.032. Epub 2021 Dec 2. PMID 34864158